CLINICAL TRIAL: NCT06351423
Title: The Effectiveness of MIND Diet and Forest Bathing on Reducing Psychological Stress Among Older Chinese: A Pilot Randomized Controlled Trial
Brief Title: The Effectiveness of MIND Diet and Forest Bathing on Stress Reduction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE-NHS2023/03
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-02

CONDITIONS: Anxiety; Depression; Stress; Psychological Stress
Keywords: MIND diet; Mediterranean-DASH Intervention for Neurodegenerative Delay; FB; Forest Bathing
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress, Psychological | interventions — Forest Therapy

STUDY DESIGN:
Intervention Model Description: a 3-arm randomized controlled study in a parallel design. Eligible participants will be randomly assigned into 3 interventions: (1) FB-MIND, (2) FB and (3) routine care-control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MIND Diet and Forest Bathing (MIND-FB) (Experimental): In this arm, participants will receive both the MIND diet and Forest Bathing (FB) intervention.
  Interventions: Behavioral: Forest Bathing (FB); Behavioral: MIND diet
- Forest bathing (FB) (Active Comparator): In this arm, participants will receive Forest Bathing intervention only.
  Interventions: Behavioral: Forest Bathing (FB)
- routine care group (No Intervention): The routine care group will be instructed to perform daily activities as usual and will receive a health talk and be given pamphlets about tips on maintaining mental well-being.

INTERVENTIONS:
Behavioral: Forest Bathing (FB) — The forest bathing (FB) intervention will be comprised of four 2-hour sessions held in a country park on four consecutive weekends during the daytime. The FB sessions will cover 1-2 kilometers per forest visit. Participants will convene at the country park entrance. An FB guide will provide a briefing and commence the forest trip. Following 20 minutes for participants to slow down and share their experiences, they will be invited to mindfully center themselves using their five senses for another 20 minutes. Subsequently, the participants will be afforded 20 minutes to wander along a designated forest path, followed by another 20 minutes during which they will be encouraged to stroll in a designated area to help foster a deep connection with the forest.
  Participants will have a 20-minute interval between each activity to share their experiences. A tea ceremony will be held at the end of each FB session.
  Arms: Forest bathing (FB); MIND Diet and Forest Bathing (MIND-FB)
Behavioral: MIND diet — The participants will undertake four three-month nutrition programmes consisting of four nutrition counselling sessions in an activity room at each participating community centre. All intervention sessions will be conducted by a registered nutritionist. In the nutrition sessions, the participants will learn to modify their diet to meet the MIND diet guidelines. The MIND diet promotes 10 healthy food groups and limits five unhealthy food groups (Morris et al., 2015a; Arjmand et al., 2022). As a reference, a 7-day sample menu will be provided which meets the required number of servings per day.
  Arms: MIND Diet and Forest Bathing (MIND-FB)

SUMMARY:
This clinical trial aims to explore the effectiveness of the Mediterranean DASH Intervention for Neurodegenerative Delay (MIND) diet and Forest Bathing (FB) in reducing psychological stress among older Chinese individuals. The main questions it aims to answer are:

1. what is the effect of FB on stress reduction
2. what is the effect of MIND on stress reduction

Participants of the MIND-FB group will participate will receive

1. FB: a two-hour FB session on four consecutive weekends in a country park,
2. MIND: four nutrition sessions, and adhere to the MIND diet for 12 weeks

Researchers will compare the FB and routine care groups to compare the effectiveness of MIND and FB in reducing psychological stress.

DETAILED DESCRIPTION:
This project is a pilot study to examine the effectiveness of Mediterranean DASH Intervention for Neurodegenerative Delay (MIND) Diet and Forest Bathing (FB) on reducing psychological stress. In recent years, mental health has become an increasingly important issue in Hong Kong. More people in Hong Kong are seeking help for mental health issues such as anxiety, depression, and stress. A 2020-2022 survey found that 1.2% of individuals aged 15 or above reported depression and 0.9% reported anxiety. Females had higher prevalence rates than males, and individuals aged 55-64 had the highest rates of depression (1.7%) and anxiety (15%). Conventional treatments have not been sufficient in managing or addressing chronic stress in individuals. Several factors including dietary intake and forest visits have been reported to be associated with psychological health. Research suggested that the MIND diets anti-inflammatory and pro-inflammatory components may reduce anxiety and depression, and forest bathing (FB) can reduce physiological and psychological stress by decreasing sympathetic nervous system activity and having a restorative effect. However, it is unclear if these approaches are effective for older adults with mild to moderate levels of psychological stress, particularly in the Chinese population. Additionally, there is a gap in the literature regarding the relationship between the MIND diet and psychological stress among the Chinese population. Therefore, it is important to investigate the potential impact of the MIND diet and forest bathing on psychological stress among older Chinese individuals.

The objectives of this study will be to:

1. examine and compare the therapeutic effects of the MIND-FB, FB and routine care on psychological stress (emotional states) and physiological stress (blood pressure and salivary cortisol level) at 4 weeks.
2. examine and compare the sustained effects of the MIND-FB, FB and routine care on these psychological and physiological stress at 12 weeks.
3. examine the therapeutic effect of the MIND-FB, FB and routine care by controlling for other individual characteristics (demographic and lifestyle characteristics, health history and current medication use).

In the short term, the study will benefit participants by providing them with either the MIND diet and forest bathing intervention or routine care, which is expected to reduce the level of psychological stress. The study results will be published in international peer-reviewed journals and presented at conferences. In the medium term, the project will offer evidence for local healthcare providers on the use of similar therapies for adults with psychological stress.

Introduction

Psychological Stress has been defined as a state of mental strain, distress, or anxiety, resulting from various challenging circumstances or events. In recent years, the coronavirus disease 2019 (COVID-19) pandemic has significantly impacted mental health worldwide, with notable increases in the prevalence of anxiety and depression, according to a scientific brief published by the World Health Organization. The brief also indicated that young people, women, and individuals with chronic diseases were at higher risk of experiencing heightened levels of stress, anxiety, and depression. In Hong Kong, in addition to the impact of the pandemic, individuals face high levels of stress and pressure in daily living, such as high cost of living, competitive work environment, and family relationships, which can result in burnout among individuals.

The benefits of the MIND diet in promoting mental health

The Mediterranean - Dietary Approaches to Stop Hypertension (DASH) Intervention for Neurodegenerative Delay (MIND) diet combines the Mediterranean and DASH diets and focuses on ten brain-healthy foods while restricting five detrimental food groups. A review study suggested that the diet might positively impact older adults' mental health due to the anti-inflammatory and pro-inflammatory properties of its components. Specific nutrients, such as long-chain n-3 fatty acids in fish and flavonoids in berries and green leafy vegetables, exhibited antioxidant and anti-inflammatory properties that inhibited amyloid-beta (Aβ) formation, which could cause brain atrophy. Limiting the intake of certain foods, such as butter, margarine, pastries, sweets, saturated fats, and trans-fats, could enhance blood-brain barrier function and mitigate Aβ aggregation. These mechanisms may have a direct impact on brain health and indirectly affect psychological health.

Several recent studies have examined the relationship between adherence to the MIND diet and mental health outcomes. One case-control study found that high adherence to the MIND diet was associated with lower anxiety scores (OR = 0.03) and significantly reduced severity of anxiety disorders (β=-3.63, p<0.001). Another cross-sectional study found that the MIND diet was significantly associated with lower odds of depression (OR=0.62) and anxiety (OR=0.61), but not psychological stress (OR=0.57). However, a cohort study did not find a significant association between MIND diet adherence and incident depression but did find reduced depression risk with the consumption of fruits, and nuts, and avoidance of fast or fried foods. Additionally, another cohort study found that the highest adherence group to the MIND diet had lower rates of depressive symptoms over time compared to the low adherence group.

The effectiveness of FB in promoting mental health

In recent years, the Japanese, Korean, and Taiwanese governments have promoted forest bathing as a therapeutic practice for urban residents. This practice involves intentional exposure to forested areas within the city to promote relaxation and well-being. Forest bathing, also known as Shinrinyoku in Japan, is a sensory experience that entails immersing oneself in natural surroundings and mindfully engaging all five senses. Theories, such as Kaplan and Kaplan's Attention Restoration Theory (ART) and Ulrich's Psycho-evolutionary Stress Reduction Theory (PET), suggested that exposure to natural environments could promote positive mood, reduce stress, restore cognitive resources, and improve mental functioning. Empirical studies have found that forest bathing has a direct effect on decreasing sympathetic nervous system activity and stress hormone levels, leading to a relaxed state. Scientific literature reviews have suggested the therapeutic effect of forest bathing on stress-related disorders, including depression, anxiety, attention deficit and hyperactivity disorders (ADHD), and stress. Therefore, forest bathing is considered a useful practice for reducing symptoms of stress and promoting relaxation and well-being.

The research team conducted a pilot randomized controlled trial (RCT) to test the therapeutic effect in three groups (the MIND diet plus FB (MIND-FB) group, the MIND group, and the control group) of older Chinese adults with hypertension. The MIND-FB group showed significant decreases in the score of state (-5.28) and trait anxiety level (-4.28), total emotional state (-6.28), tension-anxiety (-2.2), fatigue (-1.4), anger (-1.24) and confusion (-1.28) after the 4 weeks of intervention. However, it is unclear if these approaches are effective for older adults with mild to moderate levels of psychological stress, particularly in the Chinese population in reducing psychological and physiological stress. Additionally, there is a gap in the literature regarding the relationship between the MIND diet and psychological stress among the Chinese population. Further study is needed to investigate the potential impact of the MIND diet and forest bathing on psychological stress among older Chinese individuals. This randomized controlled trial will target older individuals between the ages of 50 and 75 who are at higher risk of mental illness and will investigate the effectiveness of the MIND diet and forest bathing in reducing psychological and physiological stress. We hypothesise that both interventions will offer significant mental health benefits to older Chinese individuals, with a greater reduction in psychological stress compared to physiological stress.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity, and
* able to speak and understand Cantonese, and
* the Chinese version of the DASS-21 stress subscale score larger than or equal to 8, and smaller than or equal to 12; or
* the Chinese version of the DASS-21 anxiety subscale score larger than or equal to 4, and smaller than or equal to 7, or
* the Chinese version of the DASS-21 depression subscale score larger than or equal to 5, and smaller than or equal to 10.

Exclusion Criteria:

* kidney disease and chronic obstructive pulmonary disease that is poorly controlled
* known allergies to berries, nuts, fish or olive oil
* known to mental health services
* those who participated in any relaxation or dietary programme in the past 3 months and those who anticipate joining such a programme shortly
* those who are unable to walk independently

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-03 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Emotional states | The outcome measures will be evaluated at three time points: baseline assessment (T0), immediately after the fourth session (T1), and 12 weeks following the intervention (T2) at the participating community center.
  Emotional states are measured using self-reported Chinese questionaries of depression, anxiety and stress scale -21 items (DASS-21) with alpha coefficient ranging from 0.79 to 0.83 (Cao et al., 2023).

SECONDARY OUTCOMES:
Systolic Blood Pressure (SBP) | The outcome measures will be evaluated at three time points: baseline assessment (T0), immediately after the fourth session (T1), and 12 weeks following the intervention (T2) at the participating community center.
  SBP will be determined using a validated digital automatic sphygmomanometer. BP was measured twice in a sitting position after resting for at least 10-15 min and based on the mean of two measurements of a participant.
Salivary Cortisol | The outcome measures will be evaluated at three time points: baseline assessment (T0), immediately after the fourth session (T1), and 12 weeks following the intervention (T2) at the participating community center.
  The salivary cortisol will be detected by eNano Health's saliva-based P4 Test service. Each participant will be provided with a P4 test kit to collect saliva. The saliva will be collected by placing the test cassette under the tongue for about two minutes. The collected samples were then sent to a lab for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Ling Ngai Tung, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
I would share all individual participant data (IPD) that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication.
Access Criteria: Investigators whose proposed research has received approval from the Institutional Review Boards (IRB).

REFERENCES:
- [Background] Yau KY, Law PS, Wong CN. Cardiac and Mental Benefits of Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet plus Forest Bathing (FB) versus MIND Diet among Older Chinese Adults: A Randomized Controlled Pilot Study. Int J Environ Res Public Health. 2022 Nov 8;19(22):14665. doi: 10.3390/ijerph192214665. PMID 36429384
- [Background] undefined
- [Background] Lee I, Choi H, Bang KS, Kim S, Song M, Lee B. Effects of Forest Therapy on Depressive Symptoms among Adults: A Systematic Review. Int J Environ Res Public Health. 2017 Mar 20;14(3):321. doi: 10.3390/ijerph14030321. PMID 28335541
- [Background] Fresan U, Bes-Rastrollo M, Segovia-Siapco G, Sanchez-Villegas A, Lahortiga F, de la Rosa PA, Martinez-Gonzalez MA. Does the MIND diet decrease depression risk? A comparison with Mediterranean diet in the SUN cohort. Eur J Nutr. 2019 Apr;58(3):1271-1282. doi: 10.1007/s00394-018-1653-x. Epub 2018 Mar 7. PMID 29516224
- [Background] Cherian L, Wang Y, Holland T, Agarwal P, Aggarwal N, Morris MC. DASH and Mediterranean-Dash Intervention for Neurodegenerative Delay (MIND) Diets Are Associated With Fewer Depressive Symptoms Over Time. J Gerontol A Biol Sci Med Sci. 2021 Jan 1;76(1):151-156. doi: 10.1093/gerona/glaa044. PMID 32080745
- [Background] Barkhordari R, Namayandeh M, Mirzaei M, Sohouli MH, Hosseinzadeh M. The relation between MIND diet with psychological disorders and psychological stress among Iranian adults. BMC Psychiatry. 2022 Jul 25;22(1):496. doi: 10.1186/s12888-022-04128-2. PMID 35879688